CLINICAL TRIAL: NCT01454284
Title: The Impact of LY2605541 Versus Insulin Glargine for Patients With Type 1 Diabetes Mellitus Treated With Preprandial Insulin Lispro: a Double-Blind, Randomized, 52-week Study
Brief Title: A Study in Participants With Type I Diabetes Mellitus
Acronym: IMAGINE 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12147; I2R-MC-BIAO (Other: Eli Lilly and Company); 2011-001253-82 (EudraCT Number)
Record Dates: First submitted 2011-10-14; First posted 2011-10-18 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine; LY2605541; Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LY2605541 + Insulin Lispro (Experimental): LY2605541 titrated based on blood glucose readings, administered subcutaneously (SC) once daily at bedtime for 52 weeks in combination with Insulin Lispro. Insulin Lispro titrated based on blood glucose readings, administered SC at meal times for 52 weeks.
  Interventions: Drug: LY2605541; Drug: Insulin Lispro
- Glargine + Insulin Lispro (Active Comparator): Glargine dose titrated based on blood glucose readings, administered SC once daily at bedtime for 52 weeks in combination with Insulin Lispro. Insulin Lispro dose titrated based on blood glucose readings, administered SC at meal times for 52 weeks.
  Interventions: Drug: Glargine; Drug: Insulin Lispro

INTERVENTIONS:
Drug: Glargine
  Arms: Glargine + Insulin Lispro
Drug: LY2605541
  Arms: LY2605541 + Insulin Lispro
Drug: Insulin Lispro
  Other Names: LY275585; Humalog

SUMMARY:
The purpose of this study is:

* To compare blood sugar control on LY2605541 with insulin glargine after 52 weeks of treatment.
* To compare the rate of nocturnal low blood sugar episodes on LY2605541 with insulin glargine during 52 weeks of treatment.
* To compare the number of participants on LY2605541 reaching blood sugar targets without low blood sugar episodes at night to those taking insulin glargine after 52 weeks of treatment.
* To compare the rate of low blood sugar episodes on LY2605541 with insulin glargine during 52 weeks of treatment

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for at least 1 year
* HbA1c value less than 12 percent according to the central laboratory at screening
* Body mass index of less than or equal to 35.0 kilograms per square meter (kg/m^2)
* Have been treated for at least 90 days prior to screening with

  * insulin detemir, insulin glargine, or Neutral Protamine Hagedorn (NPH) in combination with pre-meal insulin, or
  * self-mixed or pre-mixed insulin regimens with any basal and bolus insulin combination administered at least twice daily, or
  * continuous SC insulin infusion therapy
* Women who are not breast feeding and test negative for pregnancy before receiving treatment and agree to use reliable birth control until 2 weeks after last treatment with study drug
* Are capable and willing to adhere to multiple daily injections, inject with a vial and syringe and prefilled pen and perform self-monitored blood glucose (SMBG) readings and record keeping

Exclusion Criteria:

* Are using twice daily insulin glargine having been inadequately controlled on single daily dose of glargine prior to screening
* Excessive insulin resistance defined as having received a total daily dose of insulin greater than 1.5 units per kilogram (U/kg) at the time of randomization
* Receiving any oral or injectable medication (other than insulins or metformin for treatment of polycystic ovarian disease) intended for the treatment of diabetes mellitus in the 90 days prior to screening
* Lipid lowering medications:

  * are using niacin preparations as lipid lowering medication and/or bile acid sequestrants within 90 days prior to screening; or,
  * are using lipid lowering medication at a dose that has not been stable for 90 days or more prior to screening
* Have fasting hypertriglyceridemia (defined as greater than 4.5 millimoles per liter [mmol/L], greater than 400 milligrams per deciliter [mg/dL]) at screening, as determined by the central laboratory.
* Have had more than 1 episode of severe hypoglycemia (defined as requiring assistance due to neurologically disabling hypoglycemia) within 6 months prior to screening
* Have had 2 or more emergency room visits or hospitalizations due to poor glucose control within 6 months prior to screening
* Have cardiac disease with functional status that is New York Heart Association Class III or IV
* Have a history of renal transplantation or are currently receiving renal dialysis or have serum creatinine greater than 2.5 mg/dL
* Have obvious clinical signs or symptoms of liver disease (excluding non-alcoholic fatty liver disease [NAFLD]), acute or chronic hepatitis, non-alcoholic steatohepatitis (NASH), or elevated liver enzyme measurements as indicated below:

  * total bilirubin 2 times or more than the upper limit of normal (ULN) as defined by the central laboratory, or
  * alanine aminotransferase (ALT)/(serum glutamic pyruvic transaminase (SGPT) more than 2.5 times ULN as defined by the central laboratory, or
  * aspartate aminotransferase (AST)/(serum glutamic oxaloacetic transaminase (SGOT) more than 2.5 times ULN as defined by the central laboratory
* Have active or untreated malignancy, have been in remission from clinically significant malignancy (other than basal cell or squamous cell skin cancer) for less than 5 years, or are at increased risk for developing cancer or a recurrence of cancer
* Diagnosed clinically significant diabetic autonomic neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1114 (Actual)
Dates: Start 2012-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (117):
- United States (47):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Mesa, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lancaster, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tustin, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aurora, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Longmont, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bradenton, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hollywood, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Port Richey, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roswell, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Honolulu, Hawaii
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Des Moines, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Metairie, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eagan, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chesterfield, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Billings, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashua, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albany, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durham, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morehead City, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mentor, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eugene, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greer, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Myrtle Beach, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chattanooga, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Round Rock, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ogden, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Federal Way, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tacoma, Washington
- Australia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Merewether, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Keswick, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Box Hill, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parkville, Victoria
- Belgium (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edegem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huy
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sint-Niklaas
- Brazil (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fortaleza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto Alegre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Canada (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edmonton, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Red Deer, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halifax, Nova Scotia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oakville, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Laval, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osijek, Croatia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Copenhagen, Denmark
- France (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Rochelle
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Le Creuzot
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rouen
- Greece (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chalcis
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dublin, Ireland
- Israel (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haifa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jerusalem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Petah Tikva
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Litwinsky
- Lithuania (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jonava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaunas
- Netherlands (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dordrecht
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Groningen
- New Zealand (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Christchurch
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wellington
- Poland (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Katowice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lubin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szczecin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Štúrovo, Slovakia
- South Africa (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houghton Estate
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pretoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Somerset West
- Spain (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alcalá de Henares
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alzira
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Málaga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
- Sweden (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alingsås
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Helsingborg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huddinge
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Karlstad
- United Kingdom (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bristol, Avon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portsmouth, Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Blackburn, Lancashire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leicester, Leicestershire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Inverness, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ipswich, Suffolk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guildford, Surrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Swansea, Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glasgow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Northampton
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oxford

REFERENCES:
- [Derived] Qu Y, White RD, Ruberg SJ. Accurate Collection of Reasons for Treatment Discontinuation to Better Define Estimands in Clinical Trials. Ther Innov Regul Sci. 2023 May;57(3):521-528. doi: 10.1007/s43441-022-00491-0. Epub 2022 Dec 21. PMID 36542287
- [Derived] Sanyal A, Cusi K, Hartman ML, Zhang S, Bastyr EJ 3rd, Bue-Valleskey JM, Chang AM, Haupt A, Jacober SJ, Konrad RJ, Zhang Q, Hoogwerf BJ. Cytokeratin-18 and enhanced liver fibrosis scores in type 1 and type 2 diabetes and effects of two different insulins. J Investig Med. 2018 Mar;66(3):661-668. doi: 10.1136/jim-2017-000609. Epub 2017 Nov 21. PMID 29167192
- [Derived] Orchard TJ, Cariou B, Connelly MA, Otvos JD, Zhang S, Antalis CJ, Ivanyi T, Hoogwerf BJ. The effects of basal insulin peglispro vs. insulin glargine on lipoprotein particles by NMR and liver fat content by MRI in patients with diabetes. Cardiovasc Diabetol. 2017 Jun 6;16(1):73. doi: 10.1186/s12933-017-0555-1. PMID 28587667
- [Derived] Cusi K, Sanyal AJ, Zhang S, Hartman ML, Bue-Valleskey JM, Hoogwerf BJ, Haupt A. Non-alcoholic fatty liver disease (NAFLD) prevalence and its metabolic associations in patients with type 1 diabetes and type 2 diabetes. Diabetes Obes Metab. 2017 Nov;19(11):1630-1634. doi: 10.1111/dom.12973. Epub 2017 Jun 22. PMID 28417532

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2605541 + Insulin Lispro: Includes participants randomized to receive LY2605541 plus Insulin Lispro.
  Participant-specific dose of LY2605541 was administered subcutaneously (SC) once daily at bedtime for 52 weeks.
  Participant-specific dose of Insulin Lispro was administered SC at meal times for 52 weeks.
- Insulin Glargine + Insulin Lispro: Includes participants randomized to receive Insulin Glargine plus Insulin Lispro.
  Participant-specific dose of Insulin Glargine was administered SC once daily at bedtime for 52 weeks.
  Participant-specific dose of Insulin Lispro was administered SC at meal times for 52 weeks.
Period: Overall Study
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Started | 664 | 450
Received at Least 1 Dose of Study Drug | 663 | 449
Completed | 548 | 377
Not Completed | 116 | 73
Not completed — Adverse Event | 20 | 7
Not completed — Death | 0 | 3
Not completed — Lost to Follow-up | 13 | 8
Not completed — Protocol Violation | 9 | 6
Not completed — Withdrawal by Subject | 58 | 36
Not completed — Physician Decision | 16 | 11
Not completed — Sponsor Decision | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants.
Groups:
- LY2605541 + Insulin Lispro: Participant-specific dose of LY2605541 was administered SC once daily at bedtime for 52 weeks.
  Participant-specific dose of Insulin Lispro was administered SC at meal times for 52 weeks.
- Insulin Glargine + Insulin Lispro: Participant-specific dose of Insulin Glargine was administered SC once daily at bedtime for 52 weeks.
  Participant-specific dose of Insulin Lispro was administered SC at meal times for 52 weeks.
- Total: Total of all reporting groups
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro | Total
Number analyzed (Participants) | 664 | 450 | 1114
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.58 (13.50) | 42.28 (13.16) | 41.86 (13.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 267 | 169 | 436
  Male | 397 | 281 | 678
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 18 | 41
  Not Hispanic or Latino | 477 | 315 | 792
  Unknown or Not Reported | 164 | 117 | 281
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 15 | 14 | 29
  White | 625 | 426 | 1051
  More than one race | 15 | 6 | 21
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 343 | 229 | 572
  Slovakia | 5 | 5 | 10
  Greece | 15 | 8 | 23
  Spain | 44 | 30 | 74
  Ireland | 2 | 3 | 5
  Lithuania | 2 | 5 | 7
  Israel | 13 | 9 | 22
  United Kingdom | 38 | 25 | 63
  France | 12 | 7 | 19
  Canada | 33 | 19 | 52
  Belgium | 20 | 16 | 36
  Brazil | 19 | 11 | 30
  Poland | 51 | 33 | 84
  Croatia | 5 | 5 | 10
  Denmark | 0 | 1 | 1
  Australia | 22 | 17 | 39
  South Africa | 16 | 8 | 24
  Netherlands | 2 | 1 | 3
  New Zealand | 9 | 5 | 14
  Sweden | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c (HbA1c)
Description: HbA1c is a test that measures a participant's average blood glucose level over a 2 to 3 month timeframe. Least squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, stratification factors (country, baseline low density lipoprotein cholesterol [LDL-C] [<100 milligrams/deciliter (mg/dL) (2.6 millimoles/liter [mmol/L]) and ≥100 mg/dL (2.6 mmol/L)], baseline prior basal insulin therapy [insulin glargine/detemir/other]), visit, treatment-by-visit interaction, and baseline HbA1c as the fixed effects and participant as the random effect.
Time Frame: 52 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable HbA1c data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 648 | 444
percentage of HbA1c | 7.38 (0.03) | 7.61 (0.04)

2. Secondary Outcome: Hemoglobin A1c (HbA1c)
Description: HbA1c is a test that measures a participant's average blood glucose level over the past 2 to 3 months. LS means were calculated using MMRM adjusting for treatment, stratification factors (country, baseline LDL-C [<100 mg/dL (2.6 mmol/L) and ≥100 mg/dL (2.6 mmol/L)], baseline prior basal insulin therapy [insulin glargine/detemir/other]), visit, treatment-by-visit interaction, and baseline HbA1c as the fixed effects and participant as the random effect.
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 648 | 444
percentage of HbA1c | 7.09 (0.03) | 7.42 (0.03)

3. Secondary Outcome: Change From Baseline to 52 Weeks in HbA1c
Description: HbA1c is a test that measures a participant's average blood glucose level over a 2 to 3 month timeframe. LS means were calculated using MMRM adjusting for treatment, stratification factors (country, baseline LDL-C [<100 mg/dL (2.6 mmol/L) and ≥100 mg/dL (2.6 mmol/L)], baseline prior basal insulin therapy [insulin glargine/detemir/other]), visit, treatment-by-visit interaction, and baseline HbA1c as the fixed effects and participant as the random effect.
Time Frame: Baseline, 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 648 | 444
percentage of HbA1c | -0.46 (0.03) | -0.24 (0.04)

4. Secondary Outcome: Total Hypoglycemia Events
Description: Hypoglycemic episodes are defined as events which are associated with reported signs and symptoms of hypoglycemia and/or documented blood glucose (BG) concentrations of ≤70 mg/dL (3.9 mmol/L). Group mean rates of total hypoglycemia (per 30 days) are presented and were calculated from negative binomial regression models (number of episodes = treatment + baseline total hypoglycemia rate, with log [exposure in days/30] as an offset variable). Group mean is estimated by taking the inverse link function on individual participant covariates first and then averages over all participants.
Time Frame: Baseline through 26 weeks, Baseline through 52 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable data at both baseline and post-baseline.
Measure: Mean (Standard Error); unit: episodes/participant/30 days
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 662 | 449
episodes/participant/30 days
  Weeks 0-26 | 16.83 (0.36) | 14.66 (0.36)
  Weeks 0-52 | 15.34 (0.32) | 13.88 (0.35)

5. Secondary Outcome: Percentage of Participants With Total Hypoglycemic Events
Description: Hypoglycemic episodes are defined as events that are associated with the reported signs and symptoms of hypoglycemia and/or documented BG concentrations of ≤70 mg/dL (3.9 mmol/L). The percentage of participants was calculated by dividing the number of participants with hypoglycemic episodes by the total number of participants analyzed, multiplied by 100.
Time Frame: Baseline through 26 weeks, Baseline through 52 weeks
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 662 | 449
percentage of participants
  Weeks 0-26 | 99.1 | 99.3
  Weeks 0-52 | 99.2 | 99.3

6. Secondary Outcome: Percentage of Participants With HbA1c Equal to or Less Than 6.5% and Less Than 7.0%
Description: The percentage of participants was calculated by dividing the number of participants reaching target HbA1c by the total number of participants analyzed, multiplied by 100.
Time Frame: up to 26 weeks, up to 52 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable HbA1c data. Missing endpoints were imputed with the last observation carried forward (LOCF) method, using only post-baseline data.
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 648 | 444
percentage of participants
  HbA1c ≤6.5%, Week 26 | 29.6 | 17.8
  HbA1c ≤6.5%, Week 52 | 20.8 | 15.1
  HbA1c <7.0%, Week 26 | 45.1 | 34.5
  HbA1c <7.0%, Week 52 | 35.3 | 26.1

7. Secondary Outcome: Percentage of Participants With HbA1c Less Than 7.0% and Without Nocturnal Hypoglycemia
Description: Hypoglycemic episodes are defined as events associated with reported signs and symptoms of hypoglycemia and/or a documented blood glucose concentration of ≤70 mg/dL (3.9 mmol/L). A nocturnal hypoglycemic event occurred between bedtime and waking and between the time points of 10:00 PM and 10:00 AM. The percentage of participants was calculated by dividing the number of participants with HbA1c <7.0% without nocturnal hypoglycemia by the total number of participants analyzed, multiplied by 100.
Time Frame: up to 26 weeks, up to 52 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable data. Missing endpoints were imputed with the LOCF method, using only post-baseline data.
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 648 | 444
percentage of participants
  Week 26 | 7.1 | 1.8
  Week 52 | 4.3 | 1.1

8. Secondary Outcome: Nocturnal Hypoglycemia Rates
Description: Hypoglycemic episodes are defined as events that are associated with reported signs and symptoms of hypoglycemia and/or a documented BG concentration of ≤70 mg/dL (3.9 mmol/L). A nocturnal hypoglycemic event occurred between bedtime and waking and between the time points of 10:00 PM and 10:00 AM. Group mean rates of nocturnal hypoglycemia (per 30 days) are presented and were calculated from negative binomial regression models (number of episodes = treatment + baseline nocturnal hypoglycemia rate, with log [exposure in days/30] as an offset variable). Group mean is estimated by taking the inverse link function on individual participant covariates first and then averages over all participants.
Time Frame: Baseline through 26 weeks, Baseline through 52 weeks
Population: as for outcome 4
Measure: Mean (Standard Error); unit: events/participant/30 days
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 662 | 449
events/participant/30 days
  Weeks 0-26 | 1.37 (0.07) | 2.70 (0.12)
  Weeks 0-52 | 1.31 (0.06) | 2.46 (0.10)

9. Secondary Outcome: Percentage of Participants With Nocturnal Hypoglycemic Events
Description: Hypoglycemic episodes are defined as events associated with the reported signs and symptoms of hypoglycemia and/or a BG concentration of ≤70 mg/dL (3.9 mmol/L). A nocturnal hypoglycemic event occurred between bedtime and waking and between the time points of 10:00 PM and 10:00 AM. The percentage of participants was calculated by dividing the number of participants with nocturnal hypoglycemic episodes by the total number of participants analyzed, multiplied by 100.
Time Frame: Baseline through 26 weeks, Baseline through 52 weeks
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 662 | 449
percentage of participants
  Weeks 0-26 | 81.7 | 94.7
  Weeks 0-52 | 87.5 | 96.2

10. Secondary Outcome: Change in Body Weight
Description: LS means were calculated using MMRM adjusting for treatment, stratification factors (baseline HbA1c [≤8.5% and >8.5%], country, baseline LDL-C [<100 mg/dL (2.6 mmol/L) and ≥100 mg/dL (2.6 mmol/L)], baseline prior basal insulin therapy [insulin glargine/detemir/other]), visit, treatment-by-visit interaction, and baseline body weight as fixed effects and participant as the random effect.
Time Frame: Baseline, 26 weeks, 52 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable body weight data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 648 | 439
kilograms (kg)
  Week 26 | -0.55 (0.14) | 0.78 (0.16)
  Week 52 | -0.61 (0.17) | 1.21 (0.20)

11. Secondary Outcome: 9 Point Self-monitored Blood Glucose (SMBG)
Description: 9-point SMBG profiles were obtained over 2 days within the week prior to Weeks 0, 4, 12, 26, 39, and 52. SMBG measurements were taken at 9 time points: pre-morning meal, 2 hours post-morning meal, pre-midday meal, 2 hours post-midday meal, pre-evening meal, 2 hours post-evening meal, bedtime, at approximately 0300 hours, and the subsequent morning prior to the morning meal. LS means were calculated using MMRM adjusting for treatment, stratification factors (baseline HbA1c [≤8.5% and >8.5%], country, baseline LDL-C [<100 mg/dL (2.6 mmol/L) and ≥100 mg/dL (2.6 mmol/L)], baseline prior basal insulin therapy [insulin glargine/detemir/other]), visit, treatment-by-visit interaction, and baseline BG values as the fixed effects and participant as the random effect.
Time Frame: 26 weeks and 52 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable SMBG data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 615 | 416
mg/dL
  Pre-morning meal, Week 26 | 153.85 (2.67) | 148.91 (3.17)
  Pre-morning meal, Week 52 | 156.18 (2.75) | 155.25 (3.30)
  2 hour post-morning meal, Week 26: number analyzed (Participants) | 572 | 380
  2 hour post-morning meal, Week 26 | 164.59 (3.44) | 178.47 (4.07)
  2 hour post-morning meal, Week 52: number analyzed (Participants) | 572 | 380
  2 hour post-morning meal, Week 52 | 171.94 (3.43) | 183.35 (4.10)
  Pre-midday meal, Week 26: number analyzed (Participants) | 611 | 403
  Pre-midday meal, Week 26 | 136.70 (2.70) | 152.87 (3.22)
  Pre-midday meal, Week 52: number analyzed (Participants) | 611 | 403
  Pre-midday meal, Week 52 | 145.22 (2.87) | 158.50 (3.42)
  2 hour post-midday meal, Week 26: number analyzed (Participants) | 579 | 379
  2 hour post-midday meal, Week 26 | 150.66 (3.32) | 164.47 (3.94)
  2 hour post-midday meal, Week 52: number analyzed (Participants) | 579 | 379
  2 hour post-midday meal, Week 52 | 156.92 (3.73) | 172.61 (4.42)
  Pre-evening meal, Week 26: number analyzed (Participants) | 603 | 407
  Pre-evening meal, Week 26 | 155.38 (3.13) | 176.50 (3.73)
  Pre-evening meal, Week 52: number analyzed (Participants) | 603 | 407
  Pre-evening meal, Week 52 | 153.30 (3.21) | 170.83 (3.79)
  2 hour post-evening meal, Week 26: number analyzed (Participants) | 559 | 373
  2 hour post-evening meal, Week 26 | 160.50 (3.85) | 181.18 (4.54)
  2 hour post-evening meal, Week 52: number analyzed (Participants) | 559 | 373
  2 hour post-evening meal, Week 52 | 169.61 (4.19) | 184.19 (4.99)
  Bedtime, Week 26: number analyzed (Participants) | 578 | 382
  Bedtime, Week 26 | 163.90 (3.24) | 180.97 (3.84)
  Bedtime, Week 52: number analyzed (Participants) | 578 | 382
  Bedtime, Week 52 | 168.04 (3.58) | 187.09 (4.30)
  0300 Hours, Week 26: number analyzed (Participants) | 529 | 347
  0300 Hours, Week 26 | 169.64 (3.69) | 163.09 (4.39)
  0300 Hours, Week 52: number analyzed (Participants) | 529 | 347
  0300 Hours, Week 52 | 168.72 (3.94) | 174.11 (4.72)
  Pre-morning meal next day, Week 26: number analyzed (Participants) | 583 | 403
  Pre-morning meal next day, Week 26 | 150.04 (2.76) | 145.77 (3.23)
  Pre-morning meal next day, Week 52: number analyzed (Participants) | 583 | 403
  Pre-morning meal next day, Week 52 | 151.22 (2.70) | 149.56 (3.20)

12. Secondary Outcome: Fasting Serum Glucose (by Laboratory Measurement)
Description: Fasting serum glucose (FSG) is measured in blood before the morning meal. LS means were calculated using MMRM adjusting for treatment, stratification factors (baseline HbA1c [≤8.5% and >8.5%], country, baseline LDL-C [<100 mg/dL (2.6 mmol/L) and ≥100 mg/dL (2.6 mmol/L)], baseline prior basal insulin therapy [insulin glargine/detemir/other]), visit, treatment-by-visit interaction, and baseline HbA1c as the fixed effects and participant as the random effect.
Time Frame: 26 weeks and 52 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable FSG data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 646 | 443
mg/dL
  Week 26 | 139.76 (2.75) | 155.23 (3.25)
  Week 52 | 142.02 (2.95) | 171.67 (3.48)

13. Secondary Outcome: Fasting Blood Glucose (by Participant Self Monitored Blood Glucose Readings)
Description: Fasting blood glucose (FBG) was measured by SMBG pre-morning meal. LS means were calculated using MMRM adjusting for treatment, stratification factors (baseline HbA1c [≤8.5% and >8.5%], country, baseline LDL-C [<100 mg/dL (2.6 mmol/L) and ≥100 mg/dL (2.6 mmol/L)], baseline prior basal insulin therapy [insulin glargine/detemir/other]), visit, treatment-by-visit interaction, and baseline FBG as the fixed effects and participant as the random effect.
Time Frame: 26 weeks and 52 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable FBG data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 643 | 441
mg/dL
  Week 26 | 154.84 (1.96) | 151.46 (2.31)
  Week 52 | 159.85 (2.02) | 153.09 (2.39)

14. Secondary Outcome: Intra-participant Variability of Fasting Blood Glucose (FBG)
Description: FBG was measured by SMBG. Between-day glucose variability is measured by the standard deviation (SD) of FBG. LS means were calculated using MMRM adjusting for treatment, stratification factors (baseline HbA1c [≤8.5% and >8.5%], country, baseline LDL-C [<100 mg/dL (2.6 mmol/L) and ≥100 mg/dL (2.6 mmol/L)], baseline prior basal insulin therapy [insulin glargine/detemir/other]), visit, treatment-by-visit interaction, and baseline SD of FBG as the fixed effects and participant as the random effect.
Time Frame: 26 weeks and 52 weeks
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 639 | 437
mg/dL
  Week 26 | 51.70 (1.22) | 64.73 (1.44)
  Week 52 | 53.97 (1.24) | 63.11 (1.46)

15. Secondary Outcome: 0300 Hours Blood Glucose (BG) to Fasting BG Excursion
Description: Results of a 0300-hour to pre-morning meal (FBG) excursion are presented (only excursions within a single SMBG profile are included). LS means were calculated using MMRM adjusting for treatment, stratification factors (baseline HbA1c [≤8.5% and >8.5%], country, baseline LDL-C [<100 mg/dL (2.6 mmol/L) and ≥100 mg/dL (2.6 mmol/L)], baseline prior basal insulin therapy [insulin glargine/detemir/other]), visit, treatment-by-visit interaction, and baseline excursion as the fixed effects and participant as the random effect.
Time Frame: 26 weeks and 52 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable SMBG data at baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 498 | 332
mg/dL
  Week 26 | -25.49 (3.96) | -16.44 (4.72)
  Week 52 | -23.36 (4.10) | -29.01 (4.87)

16. Secondary Outcome: Triglycerides, Low Density Lipoprotein Cholesterol (LDL-C), High Density Lipoprotein Cholesterol (HDL-C), and Total Cholesterol
Description: Concentrations of cholesterol, HDL-C, and LDL-C, and triglycerides are presented. LS means were calculated using MMRM adjusting for stratification factors (baseline HbA1c [≤8.5% and >8.5%], country, LDL-C [<100 mg/dL (2.6 mmol/L) and ≥100 mg/dL (2.6 mmol/L), except for the LDL-C outcome variable], prior basal insulin therapy [insulin glargine/detemir/other]), visit, treatment, treatment-by-visit interaction, and baseline value of corresponding lipid outcome variable as the fixed effects and participant as a random effect.
Time Frame: 26 weeks and 52 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable lipid data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 650 | 446
mg/dL
  Cholesterol, Week 26 | 185.51 (1.09) | 179.30 (1.29)
  Cholesterol, Week 52 | 184.66 (1.13) | 178.13 (1.34)
  HDL-C, Week 26 | 58.44 (0.39) | 61.52 (0.46)
  HDL-C, Week 52 | 58.13 (0.39) | 59.52 (0.46)
  LDL-C, Week 26 | 106.25 (0.90) | 100.90 (1.07)
  LDL-C, Week 52 | 105.80 (0.96) | 101.20 (1.14)
  Triglycerides, Week 26 | 105.26 (2.30) | 85.11 (2.73)
  Triglycerides, Week 52 | 104.84 (2.17) | 88.12 (2.57)

17. Secondary Outcome: Percentage of Participants With Change in Anti-LY2605541 Antibodies
Description: The percentage of participants with anti-LY2605541 treatment-emergent antibody response (TEAR) is summarized. TEAR is defined as change from baseline to post-baseline in the anti-LY2605541 antibody level either from undetectable to detectable, or from detectable to the value with at least 130% relative increase from baseline.
Time Frame: 26 weeks, 52 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable anti-LY2605541 antibody data at baseline and post-baseline.
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 556 | 399
percentage of participants
  Week 26 | 30.2 | 14.0
  Week 52: number analyzed (Participants) | 509 | 363
  Week 52 | 32.8 | 10.2

18. Secondary Outcome: Basal, Meal Time, and Total Insulin Dose Per Body Weight
Description: Basal insulin dose, meal-time insulin dose (short-acting bolus dose), and total insulin dose were calculated based on the dose during the last 7 days prior to the post-treatment visit or last 3 days prior to the randomization visit. LS means were calculated using a constrained Longitudinal Data Analysis (cLDA) model adjusting for indicator variables of each treatment group at each postbaseline visit and stratification variables (baseline HbA1c [≤8.5% and> 8.5%], country, baseline LDL-C [<100 mg/dL (2.6 mmol/L) and ≥100 mg/dL (2.6 mmol/L)], and baseline prior basal insulin therapy [insulin glargine/detemir/ other]) as fixed effects.
Time Frame: 26 weeks and 52 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable insulin dose data.
Measure: Least Squares Mean (Standard Error); unit: units/weight/day
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 551 | 392
units/weight/day
  Basal insulin, Week 26: number analyzed (Participants) | 527 | 374
  Basal insulin, Week 26 | 0.46 (0.01) | 0.35 (0.01)
  Basal insulin, Week 52: number analyzed (Participants) | 508 | 367
  Basal insulin, Week 52 | 0.47 (0.01) | 0.35 (0.01)
  Meal time insulin, Week 26: number analyzed (Participants) | 542 | 388
  Meal time insulin, Week 26 | 0.32 (0.01) | 0.44 (0.01)
  Meal time insulin, Week 52: number analyzed (Participants) | 490 | 352
  Meal time insulin, Week 52 | 0.33 (0.01) | 0.43 (0.01)
  Total insulin, Week 26 | 0.75 (0.01) | 0.77 (0.01)
  Total insulin, Week 52: number analyzed (Participants) | 509 | 369
  Total insulin, Week 52 | 0.78 (0.01) | 0.77 (0.02)

19. Secondary Outcome: Insulin Treatment Satisfaction Questionnaire
Description: Insulin Treatment Satisfaction Questionnaire (ITSQ) is a validated measure containing 22 items that assess treatment satisfaction for participants with diabetes and on insulin. The questionnaire measures satisfaction from the following 5 domains: Convenience of Regimen, Lifestyle Flexibility, Glycemic Control, Hypoglycemic Control, and Insulin Delivery Device. Data are transformed to a scale of 0-100, where higher scores indicate better treatment satisfaction. LS means were calculated using an ANCOVA model adjusting for treatment, baseline HbA1c (≤8.5% and >8.5%), country, and baseline prior basal insulin therapy (insulin glargine/detemir/other) as fixed effects and baseline ITSQ scores as a covariate.
Time Frame: up to 52 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable ITSQ data at both baseline and post-baseline. Missing endpoints were imputed with the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 561 | 406
units on a scale | 73.60 (0.57) | 72.92 (0.67)

20. Secondary Outcome: European Quality of Life -5 Dimension (EQ-5D-3L)
Description: The EQ-5D-3L is a generic, multidimensional, health-related, quality-of-life instrument. The profile allows participants to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression using a three-level scale of 1-3 (no problem, some problems, and extreme problems). These combinations of attributes are converted into a weighted health-state Index Score according to the United States population-based algorithm. Scores range from -0.11 to 1.0, where a score of 1.0 indicates perfect health. LS means were calculated using an ANCOVA adjusting for treatment, baseline HbA1c (≤8.5% and >8.5%), country, baseline prior basal insulin therapy (insulin glargine/detemir/other), and baseline EQ-5D-3L score as covariates.
Time Frame: up to 52 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable EQ-5D-3L data at both baseline and post-baseline. Missing endpoints were imputed with the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 566 | 406
units on a scale | 0.91 (0.00) | 0.92 (0.01)

21. Secondary Outcome: Adult Low Blood Sugar Survey
Description: Low Blood Sugar Survey (LBSS) (also referenced as Hypoglycemia Fear Survey - II [HFS-II]) is a questionnaire that measures 1) behaviors to avoid hypoglycemia and its negative consequences (15 items) and 2) worries about hypoglycemia and its negative consequences (18 items). Responses are made on a 5-point Likert-type scale where 0 = Never and 4 = Always. Total score is the sum of all items (range 0-132). Higher total scores reflect greater fear of hypoglycemia. LS means were calculated using MMRM adjusting for treatment, baseline HbA1c (≤8.5% and >8.5%), country, baseline prior basal insulin therapy (insulin glargine/detemir/other), visit, treatment-by-visit interaction, and baseline LBSS score as the fixed effects and participant as the random effect.
Time Frame: 26 weeks and 52 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable LBSS data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 657 | 447
units on a scale
  Week 26 | 29.48 (0.55) | 29.12 (0.65)
  Week 52 | 30.43 (0.59) | 29.27 (0.70)

22. Secondary Outcome: Rapid Assessment of Physical Activity (RAPA)
Description: The RAPA questionnaire assesses the level and intensity of physical activity of adult participants. It contains 2 subscales: RAPA 1 (Aerobic) and RAPA 2 (Strength and Flexibility). RAPA 1 contains 7 questions regarding the participant's amount and intensity of physical activity, allowing each participant's aerobic activity level to be categorized as sedentary, underactive, light activity, regular underactive, or active. RAPA 2 contains 2 questions regarding participants' physical activities that increase strength and improve flexibility. Each participant's strength and flexibility activity level is then categorized as neither strength nor flexibility activity, either strength or flexibility activity (not both), both strength and flexibility activity. The percentage of participants in each RAPA 1/2 category is presented and was calculated by dividing the number of participants in each RAPA 1/2 category by the total number of participants analyzed, multiplied by 100.
Time Frame: 52 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable RAPA data.
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 367 | 254
percentage of participants
  RAPA 1, Sedentary: number analyzed (Participants) | 364 | 249
  RAPA 1, Sedentary | 1.1 | 1.2
  RAPA 1, Underactive: number analyzed (Participants) | 364 | 249
  RAPA 1, Underactive | 3.8 | 4.8
  RAPA 1, Light activity: number analyzed (Participants) | 364 | 249
  RAPA 1, Light activity | 13.7 | 14.5
  RAPA 1, Regular underactive: number analyzed (Participants) | 364 | 249
  RAPA 1, Regular underactive | 24.5 | 28.5
  RAPA 1, Active: number analyzed (Participants) | 364 | 249
  RAPA 1, Active | 56.9 | 51.0
  RAPA 2, Neither strength/flexibility | 39.0 | 46.9
  RAPA 2, Either strength/flexibility | 28.9 | 26.8
  RAPA 2, Both strength/flexibility | 32.2 | 26.4

ADVERSE EVENTS:
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Serious Adverse Events (participants affected / at risk) | 117/663 | 92/449
Other Adverse Events (participants affected / at risk) | 502/663 | 305/449
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2605541 + Insulin Lispro (N=663) | Insulin Glargine + Insulin Lispro (N=449)
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 2 (3)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Colitis microscopic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Abscess oral (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Gastritis viral (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Viraemia (Infections and infestations) | 1 (1) | 0 (0)
Accident at home (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (2) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (2)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 (3) | 6 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 71 (108) | 58 (95)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2)
Benign hydatidiform mole (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebellopontine angle tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/267 (0) | 1/169 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 4 (4) | 1 (1)
Transient global amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0/267 (0) | 1/169 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1/267 (1) | 0/169 (0)
Acute psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (2)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0/267 (0) | 1/169 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2605541 + Insulin Lispro (N=663) | Insulin Glargine + Insulin Lispro (N=449)
Diarrhoea (Gastrointestinal disorders) | 14 (16) | 16 (17)
Nausea (Gastrointestinal disorders) | 21 (27) | 17 (18)
Vomiting (Gastrointestinal disorders) | 20 (20) | 16 (21)
Injection site hypertrophy (General disorders) | 16 (20) | 0 (0)
Bronchitis (Infections and infestations) | 16 (17) | 12 (14)
Gastroenteritis (Infections and infestations) | 12 (15) | 11 (14)
Gastroenteritis viral (Infections and infestations) | 18 (18) | 15 (15)
Influenza (Infections and infestations) | 45 (47) | 22 (23)
Nasopharyngitis (Infections and infestations) | 105 (141) | 70 (99)
Sinusitis (Infections and infestations) | 29 (33) | 14 (19)
Upper respiratory tract infection (Infections and infestations) | 61 (76) | 40 (52)
Urinary tract infection (Infections and infestations) | 24 (28) | 15 (18)
Viral infection (Infections and infestations) | 7 (9) | 12 (12)
Alanine aminotransferase increased (Investigations) | 17 (17) | 3 (4)
Weight increased (Investigations) | 15 (16) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (15) | 10 (12)
Headache (Nervous system disorders) | 24 (37) | 14 (21)
Cough (Respiratory, thoracic and mediastinal disorders) | 31 (32) | 14 (15)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 (15) | 12 (12)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 55 (69) | 1 (1)
Hypertension (Vascular disorders) | 11 (12) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days